CLINICAL TRIAL: NCT05324748
Title: Repeated Corticosteroid Injections Around the Greater Occipital Nerve (GON) as Prophylactic Treatment in Chronic Cluster Headache
Brief Title: Repeated GON Injections in CCH
Acronym: REGON
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Rolf Fronczek, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 79665
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-02

CONDITIONS: Cluster Headache
Keywords: GON-injection
MeSH Terms: conditions — Cluster Headache | interventions — Methylprednisolone; Saline Solution

STUDY DESIGN:
Intervention Model Description: Bi-centre, randomized, double-blind, placebo-controlled retention trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Arm (Placebo Comparator)
  Interventions: Drug: Saline solution
- Intervention Arm (Experimental)
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Injection with prednisolon
  Arms: Intervention Arm
Drug: Saline solution — 0,9%
  Arms: Placebo Arm

SUMMARY:
Background:

- The effect of repeated GON-injections has never been studied in a double-blind randomized trial as a prophylactic therapy in a well-documented group of chronic patients. As such, (repeated) GON-injection has not yet found its place in current (inter)national treatment protocols for chronic cluster headache.

Objectives:

- The primary objective is to determine if repeated GON-injection result in effective control of cluster headache attacks for more days compared to placebo in chronic cluster headache.

Eligibility:

- Patients will be selected from the LUMC (Leiden University Medical Center) and CWZ (Canisius Wilhelmina Hospital) chronic cluster headache populations, diagnosed based upon the ICHD-3.

Design:

- Bi-centre, randomized, double-blind, placebo-controlled retention trial with a maximum follow-up of one year.

DETAILED DESCRIPTION:
A single injection of the greater occipital nerve (GON) with corticosteroids ('GON-injection') has been shown to be efficacious for the prophylactic treatment of cluster headache, with only mild, local side effects and often has its effect within days. It is a low-cost and safe treatment option; however, the beneficial effects are limited to weeks to months. This makes the injection suitable for episodic cluster headache, where periods with headache attacks last weeks to months. However, the effect of repeated GON-injections has never been studied in a double-blind randomized trial as a prophylactic therapy in a well-documented group of chronic patients. As such, (repeated) GON-injection has not yet found its place in current (inter)national treatment protocols for chronic cluster headache. The injection is often only used as a last-resort treatment in a very limited number of headache centres in a trial-and-error approach with a treatment interval varying between 3 and 6 months. It is, therefore, not known what chronic cluster headache patients can expect from this treatment.

Hypothesis: Repeated GON-injections are a safe, well-tolerated, convenient, and cost-effective therapy to rapidly and long-term reduce the attack frequency in chronic cluster headache.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤ 70 years
* Chronic cluster headache (International Classification of Headache Disorders - third edition; ICHD-3)
* Ictal pain must be always at the same side
* ≥4 weekly attacks of cluster headache in the prospective one-month baseline observation period
* On a stable regimen of cluster headache prophylactics for >4 weeks prior to onset of study treatment and agreeing not to increase the dose and not starting a new cluster prophylactic during the study period

Exclusion Criteria:

* Contra-indication against, or current use of, corticosteroids
* Occipital nerve stimulation (ONS)
* Use of anticoagulation medication or a known bleeding disorder
* Inability to use an electronic diary to monitor individual attacks and other items
* Other headaches if the patient cannot reliably distinguish them from attacks of cluster headache
* Current use of prophylactic medication for other headaches
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
mean number of days, from first injection until discontinuation, study participants remain using study medication (retention rate in survival curve) | 1 year

SECONDARY OUTCOMES:
Frequency of weekly cluster headache attacks vs. baseline | 1 year
Mean duration of attacks vs. baseline | 1 year
Mean severity (1-10) of attacks vs. baseline | 1 year
Proportion of study participants with >50% or 100% reduction in attack frequency vs. baseline | 1 year
Median injection interval | 1 year
Adverse events | 1 year
Ultrasound structural integrity of the greater occipital nerve | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Canisius Wilhelmina Ziekenhuis, Nijmegen